CLINICAL TRIAL: NCT04615234
Title: Towards Precision Medicine in Psychiatry: Clinical Validation of a Combinatorial Pharmacogenomic Approach.
Brief Title: Clinical Validation of a Combinatorial Pharmacogenomic Approach in Major Depressive Disorder
Acronym: PANDORA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: IRCCS Istituto Centro San Giovanni di Dio- Fatebenefratelli (Unknown)
Responsible Party: Principal Investigator, Antonio Vita, Head Department of Mental Health and Addiction Services, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: RF-2016-02361697
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: Treated with Genetic Test Guide (TGTG): Antidepressant monotherapy treatments according to good clinical practice for major depressive disorder guided with the pharmacogenomic test (PGs)
  Interventions: Device: Pharmacogenomics test (PGx)
- Control: Treated as Usual (TAU): Antidepressant monotherapy treatments according to good clinical practice for major depressive disorder.

INTERVENTIONS:
Device: Pharmacogenomics test (PGx) — The clinicians of the TGTG group patients receive the PGx test report within 48 hours and all the participants start the new treatment within 72 hours. According with both Clinical Pharmacogenetics Implementation Consortium (CPIC) and the Dutch Pharmacogenetics Working Group (DPWG) guidelines, the PGx report places the most ADs widespread in Italy, into three recommended categories: 1) "use as directed" (labelled as "Green"), 2) "use with caution" (labelled as "Yellow"), 3) "use with extreme caution" (labelled as "Red")
  Groups: Experimental: Treated with Genetic Test Guide (TGTG)

SUMMARY:
Major depressive disorder (MDD) is a common, chronic, debilitating mood disorder causing serious functional impairment and significantly decreased quality of life. Pharmacotherapy represents the first-line treatment choice; however, only about one third of patients respond to the first trial because of antidepressants ineffectiveness or side-effects. This causes suffering for patients and their families and significantly contributes to pushing up costs for healthcare services. Precision medicine in psychiatry might offer to clinicians the possibility to tailor the treatment according to the best possible evidence of effectiveness and tolerability for each subject. In this context our study aims to carry out a clinical validation of a combinatorial pharmacogenomics (PGx) test in an Italian MDD patient cohort with an advocacy license independence.

Our study is a prospective single-blind randomized controlled clinical observational trial enrolling 300 MDD patients. Patients referred to psychiatric services due to the failure and/or the onset of adverse effects of their current treatment for receiving a new antidepressant. Eligible participants with a primary diagnosis of MDD according to DSM-5 criteria and a Hamilton Depression Rating Scale (HAM-D17) with a score > 14 are randomized to TGTG group (Treated with Genetic Test Guide) or TAU group (Treated as Usual). For all subjects, buccal brush for DNA is collected. The primary outcome is the reduction in depressive symptomatology as measured by HAM-D17. The secondary outcomes involve a range of scales that assess MDD symptoms and social functioning outcomes. The assessment is performed at four timepoints: baseline and 4, 8, and 12 weeks. This project represents the first randomized controlled clinical trial in which is tested whether a non-commercial PGx test improves outcomes in a MDD naturalistic cohort. Moreover, the identification of new genetic variants associated with non-response or side effects will improve the efficacy of the test leading to a further cost-saving.

ELIGIBILITY:
Inclusion Criteria:

* A current diagnosis of unipolar depression according to Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5)
* An Hamilton Depression Rating Scale (HAMD-17) score >=14
* Caucasian ethnicity.

Exclusion Criteria:

* Cognitive impairment (Mini Mental State Examination MMSE <24)
* Neurological disorders
* Diagnosis of MDD with psychotic features, bipolar I and II disorders, schizophrenia spectrum and other psychotic disorders, obsessive-compulsive disorder, post-traumatic stress disorder
* Substance abuse in the last 3 months
* Comorbidity with personality disorders (cluster A and/or B); pregnancy
* Comorbidity with other severe medical illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MDD out-patients are voluntarily enrolling in the study. Patients referred to psychiatric services due to the failure and/or the onset of adverse effects of their current treatment for receiving a new AD.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical response | Baseline to 8 weeks
  Symptoms improvement as measured by the percent change in Hamilton Depression Rating Scale (HAMD-17). The higher the total score the more severe the depression

SECONDARY OUTCOMES:
Clinical response and remission | Baseline to 4 weeks, to 8 weeks and 12 weeks
  Response and remission rate at 4-, 8- and 12-weeks according to Hamilton Depression Rating Scale (HAMD-17). 0-7 not depressed; 8-13 mild; 14-18 moderate; 19-22 severe; >23 very severe

OTHER OUTCOMES:
Clinical response and remission self-reported | Baseline to 4 weeks, to 8 weeks and 12 weeks
  Changes in scores of depressive symptoms as measured by the Beck Depression Inventory II (BDI-II). Score on the BDI-II can range from 0 to 63 with higher scores indicating greater severity of depression
Psychosocial functioning | Baseline to 8 weeks and 12 weeks
  Changes in scores of psychosocial functioning as measured by the Mini-ICF-APP Social Functioning Scale (Mini-ICF-APP). All of items are rated using a 4-point scale, with higher ratings reflecting more severe limitations.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Mental Health and Addiction, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Minelli A, Barlati S, Vitali E, Bignotti S, Dattilo V, Tura GB, Maffioletti E, Giacopuzzi E, Santoro V, Perusi G, Cobelli C, Magri C, Bonizzato S, Bocchio-Chiavetto L, Spina E, Vita A, Gennarelli M. Clinical validation of a combinatorial PharmAcogeNomic approach in major Depressive disorder: an Observational prospective RAndomized, participant and rater-blinded, controlled trial (PANDORA trial). Trials. 2021 Dec 11;22(1):896. doi: 10.1186/s13063-021-05775-8. PMID 34895291